CLINICAL TRIAL: NCT06880666
Title: Minimally Invasive Surgical Intervention for Hirschsprung Disease: A Prospective Study on Efficacy and Long-term Functional Outcomes for Neonatal Patients
Brief Title: Minimally Invasive Surgical Intervention for Hirschsprung Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Children's Hospital, Vietnam (Other)
Responsible Party: Principal Investigator, Nguyen Thanh Quang, Principle Investigator, National Children's Hospital, Vietnam
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS50/BB - HĐĐĐ
Record Dates: First submitted 2025-03-02; First posted 2025-03-18 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Hirschsprung Disease
Keywords: Aganglionic bowel; Minimally invasive; Laparoscopic; Single incision; Pediatric; Hirschsprung
MeSH Terms: conditions — Hirschsprung Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MIS-Treated Hirschsprung Patients (2020-2024) (Experimental): Neonatal patients diagnosed with Hirschsprung's Disease, admitted to the National Children's Hospital between 2020 to 2021, and underwent Single incision laparoscopic surgery
  Interventions: Procedure: Minimally invasive laparoscopic pull-through surgery

INTERVENTIONS:
Procedure: Minimally invasive laparoscopic pull-through surgery — Conventional laparoscopic pull-through (CLP) surgery utilizes 3-5 small abdominal incisions for the placement of trocars, allowing the insertion of a laparoscopic camera and surgical instruments. After establishing pneumoperitoneum, the aganglionic segment is identified, and the colon is mobilized by dividing the lateral attachments using laparoscopic energy devices. The rectal dissection is performed circumferentially down to the level of the pelvic floor while preserving the mesenteric blood supply. A transanal approach is then used to complete the dissection, pull the mobilized bowel through the anus, and resect the aganglionic segment. A coloanal anastomosis is created, typically with absorbable sutures. Single-incision laparoscopic pull-through (SILS) follows the same principles but is performed through a single umbilical incision using a multi-port device; instruments and a camera are inserted through the same access point.

SUMMARY:
Hirschsprung's disease (HD) is one of the most common congenital conditions, with a global incidence of 1/5000 newborns; the prevalence in the Vietnamese population is even higher. The absence of enteric ganglia in the distal bowel causes intestinal obstruction and delayed meconium passage in newborns, as well as failure of normal defecation later in life. If left untreated, HD can lead to life complications such as enterocolitis and even death. Standard treatment involves surgical resection of the affected bowel segment, with minimally invasive laparoscopic techniques offering reduced postoperative complications, shorter hospital stays, and faster recovery compared to open surgery. Since 2012, the National Children Hospital has been the first institution in Vietnam to routinely use the minimally invasive surgical approach for HD. However, due to a lack of research funding and patients' financial constraints to travel to post-operative treatment centers, there has yet to be a publication addressing the long-term outcomes and associated abnormalities of all patients treated with SILS. Thus, the purpose of this study is to report on the safety, efficacy, and long-term functional outcomes and cosmesis results of minimally invasive surgeries performed on HD neonatal patients at The National Children's Hospital from 2020 to 2021, thus optimize surgical management and improve patient outcomes in a lower-middle-income country setting.

DETAILED DESCRIPTION:
Hirschsprung's disease (HD) is one of the most common congenital disorders affecting the gastrointestinal tract, with a global incidence of approximately 1 in 5,000 live births. However, studies suggest that the prevalence is notably higher in the Vietnamese population. The condition arises due to the absence of enteric ganglion cells in the distal colon, leading to a functional obstruction that prevents normal bowel motility. This defect results in delayed meconium passage in newborns, severe constipation, abdominal distension, and feeding intolerance. If left untreated, HD can progress to life-threatening complications such as Hirschsprung-associated enterocolitis (HAEC), bowel perforation, sepsis, and even death.

Surgical intervention remains the mainstay of treatment for HD, with the goal of resecting the aganglionic bowel segment and restoring normal intestinal function. Traditionally, open pull-through procedures were the standard approach, but advancements in minimally invasive surgery (MIS) have led to the widespread adoption of laparoscopic techniques. Georgeson's traditional three-port laparoscopic rectal pull-through technique, first introduced in 1995, has been widely used as the standard treatment for HD. The first case of single-incision laparoscopic assisted rectal pull-through (SILS) surgery for HD was published in 2010, in which six patients who underwent SILS all had positive outcomes and excellent cosmesis. Compared to conventional open surgery, laparoscopic approaches offer several benefits, including reduced postoperative pain, fewer wound-related complications, shorter hospital stays, improved cosmetic outcomes, and faster overall recovery. Despite the promising outcomes of minimally invasive surgical intervention, 15 years after the first reported case, only a few articles (a total of 9 articles reported in Pubmed) have been published to evaluate SILS in HD.

Since 2012, the Vietnam National Children's Hospital (NCH) has been a pioneer in the routine use of the minimally invasive surgical technique for the treatment of Hirschsprung's disease in Vietnam. However, despite over a decade of experience with this method, research on long-term outcomes in Vietnamese patients remains scarce. A major challenge has been the limited availability of research funding and the financial difficulties faced by many families, which prevent regular postoperative follow-ups and comprehensive long-term studies. As a result, there is currently no published data evaluating the long-term safety, efficacy, and potential postoperative complications associated with minimally invasive intervention for HD in this specific patient population.

The primary objective of this study is to bridge this knowledge gap by systematically analyzing the outcomes of pediatric patients who underwent minimally invasive surgical intervention for Hirschsprung's disease at NCH between 2020 and 2021. The study aims to assess key factors such as perioperative outcomes, postoperative bowel function, the incidence of complications such as anastomotic stricture or incontinence, associated abnormalities/ comorbidities, cosmesis, and quality of life improvements. By providing robust clinical evidence, this research will contribute to optimizing surgical management strategies for Hirschsprung's disease in resource-limited settings, ultimately improving patient outcomes and guiding future surgical practices in Vietnam and other LMICs.

ELIGIBILITY:
Inclusion Criteria:

* Age: From 1 to 28 days old
* Diagnosis: Hirschsprung disease was diagnosed based on clinical presentation, intraoperative frozen section biopsy, and postoperative histopathological findings showing absence of ganglion cells.
* Surgical Approach: Patients underwent SILEP through a single periumbilical incision, with no additional abdominal incisions. All surgeries were conducted by the same team, and postoperative care was provided according to a standardized protocol.
* Parents or guardians provided consent to participate in the study and committed to following the scheduled follow-up visits.

Exclusion Criteria:

* Patients exhibiting severe HAEC, bowel obstruction, or peritonitis at the time of operation
* Those with a history of failed Hirschsprung disease surgery, prior abdominal operations, or colostomy
* Individuals with contraindications to laparoscopic procedures, such as bleeding disorders or significant congenital heart defects
* Cases where parents or legal guardians refused consent for study participation

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Volume of Blood Loss | Perioperative
  The amount of blood lost during surgery will be measured in milliliters (mL) by collecting blood from suction devices, counting soaked surgical sponges, and assessing any other visible loss
Conversion to open surgery | Perioperative
  The proportion of cases in which single-incision laparoscopic surgery (SILS) could not be optimally completed and required conversion to open surgical techniques. Conversion may be necessitated by factors such as poor visualization, uncontrolled bleeding, adhesions, or patient-specific anatomical challenges. The outcome will be measured as the percentage of procedures requiring conversion during the perioperative period.
Operative time | Perioperative
  Total duration of the surgical procedure from skin incision to closure, measured in minutes.
Mortality and severe morbidity | Through study completion, an average of 4 years
  The incidence of mortality and severe postoperative complications following single-incision laparoscopic pull-through surgery. Severe morbidity includes life-threatening conditions such as sepsis, multi-organ failure, other major complications requiring intensive medical intervention, and death. This outcome will be assessed throughout the study period.
Early postoperative complications | Up to 8 weeks post-operation
  The incidence of early postoperative complications, including but not limited to bowel obstruction, surgical site infections, and Hirschsprung-associated enterocolitis (HAEC). Additional complications such as anastomotic leakage, prolonged ileus, or unexpected reoperation will also be monitored.
Rintala score | Through study completion, an average of 4 years
  The Rintala Score assesses postoperative bowel function in pediatric Hirschsprung disease (HD) patients, ranging from 0 to 20. It evaluates stool frequency, incontinence, constipation, and social continence. Scores of 18-20 indicate excellent function with normal bowel habits and no incontinence. Scores of 10-17 suggest moderate function, with occasional issues like constipation or minor incontinence. Scores below 10 reflect poor function, often requiring medical or surgical intervention.
Manchester Scar Scale | Through study completion, an average of 4 years
  The Manchester Scar Scale (MSS) evaluates the aesthetic and physical characteristics of scars, scoring from 4 to 28. It assesses scar color, contour, texture, distortion, and patient discomfort. Lower scores (4-8) indicate minimal scarring with good cosmetic outcomes. Moderate scores (9-18) suggest noticeable but acceptable scars with some textural or color irregularities. Higher scores (19-28) reflect severe scarring, often associated with significant discoloration, contour defects, or functional impairment.

SECONDARY OUTCOMES:
Associated conditions | Through study completion, an average of 4 years
  Incidence of any medical or surgical conditions identified before or after laparoscopic pull-through surgery, assessed through clinical evaluation, imaging, and diagnostic testing.

CONTACTS AND LOCATIONS:
Overall Officials: Quang T Nguyen, M.D., Principal Investigator — Department of Pediatric Surgery, The National Hospital of Pediatrics, Hanoi, Vietnam
Locations (1):
- Department of Surgery, The National Children Hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu, M., Fang, Y., Zhang, B., Lin, Y., Li, O., Bai, J., … & Wu, D. (2020). Laparoscopic-assisted soave operation for the treatment of hirschsprung disease in children: 5 years of experience.. https://doi.org/10.21203/rs.3.rs-18886/v1
- [Background] LÊ NH. ĐÁNH GIÁ KẾT QUẢ PHẪU THUẬT BỆNH GIÃN ĐẠI TRỰC TRÀNG BẨM SINH Ở NGƯỜI LỚN TẠI BỆNH VIỆN VIỆT ĐỨC. 2020
- [Background] Puri P, Nakamura H. Epidemiology and Clinical Characteristics of Hirschsprung's Disease. In: Hirschsprung's Disease and Allied Disorders
- [Background] Mayo Clinic. Hirschsprung's disease - Symptoms and causes 2021
- [Background] Georgeson KE, Robertson DJ. Laparoscopic-assisted approaches for the definitive surgery for Hirschsprung's disease. Semin Pediatr Surg. 2004 Nov;13(4):256-62. doi: 10.1053/j.sempedsurg.2004.10.013. PMID 15660319
- [Background] Zimmermann P, Martynov I, Perger L, Scholz S, Lacher M. 20 Years of Single-Incision-Pediatric-Endoscopic-Surgery: A Survey on Opinion and Experience Among International Pediatric Endosurgery Group Members. J Laparoendosc Adv Surg Tech A. 2021 Mar;31(3):348-354. doi: 10.1089/lap.2020.0797. Epub 2020 Dec 31. PMID 33395367
- [Background] Xia X, Li N, Wei J, Zhang W, Yu D, Zhu T, Feng J. Single-incision laparoscopic versus conventional laparoscopic surgery for Hirschsprung's disease: A comparison of medium-term outcomes. J Pediatr Surg. 2016 Mar;51(3):440-3. doi: 10.1016/j.jpedsurg.2015.10.051. Epub 2015 Oct 24. PMID 26611332
- [Background] Fearmonti R, Bond J, Erdmann D, Levinson H. A review of scar scales and scar measuring devices. Eplasty. 2010 Jun 21;10:e43. PMID 20596233
- [Background] Nguyen LT, Nguyen AT, Nguyen QT, Tran QA, Bui HD, Pham HD. Suspension sutures facilitate single-incision laparoscopic-assisted rectal pull-through for Hirschsprung disease. BMC Surg. 2021 May 31;21(1):274. doi: 10.1186/s12893-021-01260-w. PMID 34059040
- [Background] Ure BM, Rintala RJ, Holschneider AM. Scoring postoperative results. Anorectal Malformations Child Embryol Diagnosis, Surg Treat Follow. 2006;351-9.
- [Background] Muensterer OJ, Chong A, Hansen EN, Georgeson KE. Single-incision laparoscopic endorectal pull-through (SILEP) for hirschsprung disease. J Gastrointest Surg. 2010 Dec;14(12):1950-4. doi: 10.1007/s11605-010-1299-3. Epub 2010 Aug 18. PMID 20717739
- [Background] Amiel J, Lyonnet S. Hirschsprung disease, associated syndromes, and genetics: a review. J Med Genet. 2001 Nov;38(11):729-39. doi: 10.1136/jmg.38.11.729. PMID 11694544